CLINICAL TRIAL: NCT04425304
Title: The Effects of an Efficient Lifestyle Counseling Method on the Risks of Cardiovascular Disease in Health Care Center Patients
Brief Title: Effects of Efficient Lifestyle Counseling Method on the Risks of Cardiovascular Disease in Health Care Center Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Janne Hukkanen, Professor of Internal Medicine, University of Oulu
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Resepti-Onnikka
Record Dates: First submitted 2020-06-06; First posted 2020-06-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group counseling (Active Comparator)
  Interventions: Behavioral: Group counseling
- Group counseling + persuasive ICT support (Experimental)
  Interventions: Behavioral: Group counseling; Behavioral: Persuasive ICT support
- Intensive group counseling (Active Comparator)
  Interventions: Behavioral: Intensive group counseling
- Intensive group counseling + persuasive ICT support (Experimental)
  Interventions: Behavioral: Intensive group counseling; Behavioral: Persuasive ICT support

INTERVENTIONS:
Behavioral: Group counseling — 4 times
  Arms: Group counseling; Group counseling + persuasive ICT support
Behavioral: Intensive group counseling — 14 times
  Arms: Intensive group counseling; Intensive group counseling + persuasive ICT support
Behavioral: Persuasive ICT support — Weekly reminders for 12 months
  Arms: Group counseling + persuasive ICT support; Intensive group counseling + persuasive ICT support

SUMMARY:
The aim of the trial is to study the effect of a lifestyle change program in patients with obesity and risk of cardiovascular diseases. The main focus is to motivate and support lifestyle changes.

Two different group counseling methods (intensive and standard) with or without internet support will be compared. Thus, the patients will be randomized into four arms. Patients will be recruited from local general practice teams. The intensive lifestyle counseling consists of 12 group counseling sessions and 2 personal counseling sessions. The standard counseling consists of 4 group sessions. The internet-based counseling contains aspects of cognitive behavior therapy and persuasive design system and consists of weekly reminders, tasks, self-monitoring, and reflection.

The main outcome is the decrease in body weight. Secondary outcomes are changes in eating behavior, eating habits, components of metabolic syndrome (waist circumference, plasma lipid and glucose values), and calculated scores of cardiometabolic condition, cardiovascular risk and adiposity.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 30 to 40 kg/m2
* + 2 risk factors of cardiovascular diseases:

  * Elevated blood pressure or hypertension
  * High LDL or hypocholesterolemic drug
  * Low HDL or hypocholesterolemic drug
  * Elevated triglyceride value or hypolipidemic drug
  * Elevated glucose value or diabetes medication
  * Smoking
* Access to email and internet

Exclusion Criteria:

* Untreated hypothyroidism
* Oral corticosteroid treatment
* Pregnancy and lactation
* Angina pectoris
* Cardiac insufficiency
* Coronary Heart Disease
* Inability to speak Finnish
* Anticipated lack of compliance

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Baseline to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Janne Hukkanen, MD, PhD, Principal Investigator — University of Oulu, Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No